CLINICAL TRIAL: NCT06877130
Title: Effect of Blood Flow Restriction on Cardiovascular Function in Elderly with Metabolic Syndrome X
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Karim Mohsen Abdeltawaab, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005597
Record Dates: First submitted 2025-03-02; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Metabolic Syndrome X; Cardiovascular Problems in Elderly
Keywords: Metabolic Syndrome X; Blood Flow Restriction (BFR) Training Effects; Cardiovascular Functions in Elderly
MeSH Terms: conditions — Metabolic Syndrome | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (aerobic exercise with BFR group) (Experimental): Thirty patients will apply moderate aerobic exercise with RBF in form of a treadmill for 30 minutes for 12 weeks (3 sessions/ week).
  Interventions: Other: Aerobic exercise with BFR; Other: Aerobic training
- Group B (aerobic training group) (Active Comparator): Thirty patients will apply moderate intensity aerobic exercise without BFR for 30 minutes for 12 weeks (3 sessions/ weak).
  Interventions: Other: Aerobic training

INTERVENTIONS:
Other: Aerobic exercise with BFR — To prescribe BFR training, Systolic blood pressure (SBP) will be measured using an automated oscillometer BP device.
  Blood pressure will be measured according to the recommendations of the American Heart Association. A bilateral restriction of 50% of the measured SBP will be applied to each lower limb for the application of BFR of lower limbs using the equipment. A wide cuff (18 cm wide) will be placed in the proximal portion of the thigh (inguinal fold region) and will be inflated until the absence of the tibial artery blood pulse. Thus, a 50% restriction of SBP will be applied in both legs during lower body exercises.
  Arms: Group A (aerobic exercise with BFR group)
Other: Aerobic training — HR max = 206.9 - (0.67 x age).
  Moderate intensity aerobic exercise: the rate of heart reaches 64-76 percent of their age predicted peak hearty rate

SUMMARY:
The purpose of the study is to investigate the effect of aerobic exercise with Blood flow restriction training (BFR) on cardiovascular function and quality of life in hypertensive elderly patients.

Hypothesis There will be no significant effect of aerobic exercise with RBF on cardiovascular function and the quality of life in hypertensive elderly patients.

DETAILED DESCRIPTION:
Sixty elderly patients with metabolic syndrome X aged from 65 to 75 years old. will be selected from Al-Ahrar teaching hospital -zagazig governorate.

Study Design:

This experimental comparative control study will be performed after patients' clinical assessment who will be randomly allocated into two equal groups:

Group A (aerobic exercise with BFR group):

Thirty patients will apply moderate aerobic exercise with RBF in form of a treadmill for 30 minutes for 12 weeks (3 sessions/ week).

Group B (aerobic training group):

Thirty patients will apply moderate intensity aerobic exercise without BFR for 30 minutes for 12 weeks (3 sessions/ weak).

Equipment:

A- Evaluative Equipment:

1. Weight and height scale: (ZT-120 model, health scale made in china).
2. Sphygmomanometer: (Model Number: GT001-110/111 aneroid sphygmomanometer, Zhejiang, China)
3. Pulse oximeter: (Pulse Oximeter GRANZIA Model No: AS-304).
4. Lab investigation: using blood sample to test the following factors A- Lipid Profile: Cobas Integra 400 Plus- Switzerland. B- Apolipoprotien: Cobas Integra 400 plus -Switzerland.
5. Functional assessment:

   A-Timed Up and Go (TUG) Test The Timed Up and Go (TUG) test is a reliable, cost-effective, safe, and time-efficient way to evaluate overall functional mobility.

   B- Fatigue Assessment Scale (FAS): it is a way of measuring physical activity intensity level.
6. Quality of life assessment by using HeartQoL questionnaire

B) Treatment Equipment:

1. Treadmill, (Model Grand Fit Ac 8885- china)
2. BFR Training Therapy Occlusion Air Cuffs.

III) Procedures:

A- Evaluating Procedure:

History will be carefully taken to collect data about his general condition, physical therapy, and current medication.

The procedure of this study will be divided into the following main parts:

Preparatory procedure:

A. All medical and demographic data of subjects will be collected. B. Vital signs will be measured to ensure that all subjects are medically stable.

c. Recording data sheet: All data and information of each patient who participated in this study including name, age, address, weight, and height were recorded in the recording datasheet.

1. Weight and height:

   A valid and reliable universal height and weight scale is used to determine the subjects' height and weight. Before treatment, each patient's height- and -weight were calculated to determine their body's mass index (BMI) using the following equation: BMI=weight (Kgs) /height (m2)
2. Blood pressure monitoring by (Aneroid Sphygmomanometers) Aneroid sphygmomanometers were used to obtain a BP reading.
3. Pulse rate by Pulse oximeter:

   It is widely used to noninvasively assess arterial oxyhemoglobin saturation (SpO2) and rate of heart (HR) during rest and activity.
4. Lipid profile:

   All patients will perform laboratory lipid profile before and after the study. The three main blood levels collected to assess for dyslipidemia is (TG, HDL-C, LDL-C and T.G) after fasting for 8-12 hours. (Rosenson et al.2021).
5. apolipoprotien test: test to detect the risk of cardiovascular disease
6. Functioal assessment

   A-time up and go test:

   A sturdy armchair with a back was placed at the end of a hallway adjacent to where height and weight measures are routinely taken in the process of rooming participants.

   A piece of tape was placed on the floor 3 m away from the front edge of the chair. Patients were seated in the chair with back against the chair back, arms resting on the armrests, and given general instructions about the task, including walking at a normal rather than a rapid speed.

   The TUG required patients to stand up out of the chair, walk 3 m, turn around, walk back to the chair, and sit down. Patients were given the following instructions: "stand up on the word 'go,' walk to the tape, turn around, walk back to the chair, and sit down." The timing of the test began at the word "go," and ended when the participant was seated.

   B- Fatigue Assessment Scale (FAS) The FAS is a 10-item scale evaluating symptoms of chronic fatigue. In contrast to other similar measures the FAS treats fatigue as a unidimensional construct and does not separate its measurement into different factors. However, in order to ensure that the scale would evaluate all aspects of fatigue, developers chose items to represent both physical and mental symptoms.

   Each item of the FAS is answered using a five-point scale ranging from 1 ("never") to 5 ("always"). Items 4 and 10 are reverse scored. Total scores can range from 10, indicating the lowest level of fatigue, to 50, denoting the highest.
7. HeartQoL questionnaire. According to European Journal of Preventive Cardiology 2016 HeartQoL is a recently developed core health-related quality of life instrument for patients with coronary heart disease. The current study aims to investigate its association with patients' coronary risk profile and to provide reference values for patients with coronary heart disease (Appendix II).
8. The double product (DP): consisting of the SBP multiplied by the pulse rate (PR), is an index of myocardial oxygen consumption.
9. Mean Arterial Pressure:

The definition of mean arterial pressure (MAP) is the average arterial pressure throughout one cardiac cycle, systole, and diastole. MAP is influenced by cardiac output and systemic vascular resistance, each of which is influenced by several variables. (DeMers D et al 2023).

A common method used to estimate the MAP is the following formula:

• MAP = DP + 1/3(SP - DP)

B) Therapeutic procedure:

- Aerobic exercise training

1. Target heart rate:

   Maximum Heart Rate Formula:

   HR max = 206.9 - (0.67 x age) (Jackson et al., 2007). Moderate intensity aerobic exercise: the rate of heart reaches 64-76 percent of their age predicted peak hearty rate (American College of Sports Medicine et al. 2018).
2. Determination of BFR To prescribe BFR training, Systolic blood pressure (SBP) will be measured using an automated oscillometer BP device

Blood pressure will be measured according to the recommendations of the American Heart Association. A bilateral restriction of 50% of the measured SBP will be applied to each lower limb for the application of BFR of lower limbs using the equipment. A wide cuff (18 cm wide) will be placed in the proximal portion of the thigh (inguinal fold region) and will be inflated until the absence of the tibial artery blood pulse. Thus, a 50% restriction of SBP will be applied in both legs during lower body exercises.

ELIGIBILITY:
Inclusion Criteria:

1. sixty elderly patients.
2. Their ages will range from 60 to 70 years old.
3. Grade II Hypertensive patients (SBP 160-179 mmHg and/or DBP 100-109 mmHg)
4. Patients with dyslipidemia: at least one of the fasting lipid profile tests include the following results.

   A-Total Cholestrol more than 240 (mg/dl). B-LDL Cholestrol more than 160 (mg/dl). C-HDL Cholestrol less than 40 (mg/dl). D-Triglycerides more than 200 (mg/dl).
5. 'Body Mass Index: from 30: 40 kg/m2 calss I and II obesity.

Exclusion Criteria:

1. Severe Chest diseases (either obstructive or restrictive).
2. Clinical signs of a severe cardiac event. (eg, severe atherosclerosis, congestive heart failure),
3. Severe psychiatric or cognitive impairment, who unable to follow comment.
4. Neurological disorders affecting respiratory muscles or any muscular dystrophies (cervical disc or bulge).
5. Patients with severe self-limiting illness (e.g., cancer).
6. Peripheral artery disease in lower extremities.
7. Systolic blood pressure < 180 mmHg, diastolic blood pressure more than 110 mmHg, or resting heart rate above 120 bpm.
8. Patient with uncontrolled - diabetes.

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Weight and height measurement | Baseline (assessment).
  Weight and height are recorded, and BMI will be calculated according to the formula: BMI = Weight (Kg) / Height (m2)
Blood pressure monitoring by (Aneroid Sphygmomanometers) | Baseline (assessment), and at 12 weeks post-intervention.
  Aneroid sphygmomanometers were used to obtain a BP reading (Pickering TG et al., 2005). Virtually 100% of the values. From the aneroid-device were within the three-mm-Hg range recommended' by the Association for the Advancement of Medical instrumentation.
Pulse rate by Pulse oximeter | Baseline (assessment), and at 12 weeks post-intervention.
  It is widely used to noninvasively assess arterial oxyhemoglobin saturation (SpO2).
Lipid profile | Baseline (assessment), and at 12 weeks post-intervention.
  All patients will perform laboratory lipid profile before and after the study. The three main blood levels collected to assess for dyslipidemia is (TG, HDL-C, LDL-C and T.G) after fasting for 8-12 hours.
apolipoprotien test | Baseline (assessment), and at 12 weeks post-intervention.
  : test to detect the risk of cardiovascular disease
time up and go test | Baseline (assessment), and at 12 weeks post-intervention.
  A sturdy armchair with a back was placed at the end of a hallway adjacent to where height and weight measures are routinely taken in the process of rooming participants.
  A piece of tape was placed on the floor 3 m away from the front edge of the chair. Patients were seated in the chair with back against the chair back, arms resting on the armrests, and given general instructions about the task, including walking at a normal rather than a rapid speed.
  The TUG required patients to stand up out of the chair, walk 3 m, turn around, walk back to the chair, and sit down. Patients were given the following instructions: "stand up on the word 'go,' walk to the tape, turn around, walk back to the chair, and sit down." The timing of the test began at the word "go," and ended when the participant was seated
Fatigue Assessment Scale | Baseline (assessment), and at 12 weeks post-intervention.
  The FAS is a 10-item scale evaluating symptoms of chronic fatigue. In contrast to other similar measures the FAS treats fatigue as a unidimensional construct and does not separate its measurement into different factors. However, in order to ensure that the scale would evaluate all aspects of fatigue, developers chose items to represent both physical and mental symptoms.
  Each item of the FAS is answered using a five-point scale ranging from 1 ("never") to 5 ("always"). Items 4 and 10 are reverse scored. Total scores can range from 10, indicating the lowest level of fatigue, to 50, denoting the highest.
HeartQoL questionnaire | Baseline (assessment), and at 12 weeks post-intervention.
  According to European Journal of Preventive Cardiology 2016 HeartQoL is a recently developed core health-related quality of life instrument for patients with coronary heart disease. The current study aims to investigate its association with patients' coronary risk profile and to provide reference values for patients with coronary heart disease
The double product (DP) | Baseline (assessment), and at 12 weeks post-intervention.
  consisting of the SBP multiplied by the pulse rate (PR), is an index of myocardial oxygen consumption
Mean Arterial Pressure | Baseline (assessment), and at 12 weeks post-intervention.
  The definition of mean arterial pressure (MAP) is the average arterial pressure throughout one cardiac cycle, systole, and diastole. MAP is influenced by cardiac output and systemic vascular resistance, each of which is influenced by several variables.
  A common method used to estimate the MAP is the following formula:
  MAP = DP + 1/3(SP - DP)

CONTACTS AND LOCATIONS:
Overall Officials: Zeinab Mohamed Helmy, Professor of Physical Therapy, Study Chair — Professor of Physical Therapy for Cardiovascular / Respiratory Disorders and Geriatrics Faculty of Physical Therapy Cairo University; Ebtesam Nabil Abdel Mohsen, Lecturer of Physical Therapy, Study Director — Lecturer of Physical Therapy for Cardiovascular / Respiratory Disorders and Geriatrics Faculty of Physical Therapy Cairo University; Yasser Abdel Monem Elhendy, Professor of Internal Medicine, Study Director — Professor of Internal Medicine Faculty of Medicine Zagazig University
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No